CLINICAL TRIAL: NCT06375798
Title: Clinical Study of Breast Conserving Surgery Combined With Intraoperative Radiotherapy for Early Breast Cancer
Status: Recruiting | Type: Observational
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Cuizhi GENG, professor, Hebei Medical University Fourth Hospital
Other Study IDs: 2020137
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; HER2-negative Breast Cancer
Keywords: Breast preservation surgery; Breast cancer invasion; radiotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IORT group: The IORT group received intraoperative radiotherapy with a regimen of 50-KV-X 20Gy/1f.If the postoperative paraffin pathology of patients in the IORT group indicated positive axillary lymph nodes, the radiologist should determine whether to irradiate the whole milk and lymph nodes in the drainage area.
  Interventions: Procedure: radiotherapy
- WBI group: WBI group received whole milk external irradiation with a regimen of 50Gy/25f.If the postoperative pathology of patients in the WBI group indicated the need for chemotherapy, radiotherapy was initiated within 6 weeks after the end of chemotherapy, allowing both endocrine therapy and radiotherapy to be performed simultaneously.
  Interventions: Procedure: radiotherapy

INTERVENTIONS:
Procedure: radiotherapy — If the postoperative paraffin pathology of patients in the IORT group indicated positive axillary lymph nodes, the radiologist should determine whether to irradiate the whole milk and lymph nodes in the drainage area.If the postoperative pathology of patients in the WBI group indicated the need for chemotherapy, radiotherapy was initiated within 6 weeks after the end of chemotherapy, allowing both endocrine therapy and radiotherapy to be performed simultaneously. Clinical standard treatment plan (chemotherapy, endocrine therapy, etc.) was developed based on postoperative pathological and immunohistochemical reports.

SUMMARY:
A Single-center, open, prospective study，for analyzing the local recurrence rate, the incidence of incision complications and the aesthetic effect of intraoperative radiotherapy in early breast cancer patients after breast-conserving surgery.

DETAILED DESCRIPTION:
This is a single-center, open, prospective study. A total of 620 breast cancer patients meeting the exclusion criteria were included and assigned to the IORT group and the WBI group according to the patients' wishes. The IORT group received intraoperative radiotherapy with a regimen of 50-KF-x 20Gy/1f, and the WBI group received whole milk external irradiation with a regimen of 50Gy/25f. If the postoperative paraffin pathology of patients in the IORT group indicated positive axillary lymph nodes, the radiologist should determine whether to irradiate the whole milk and lymph nodes in the drainage area. If the postoperative pathology of patients in the WBI group indicated the need for chemotherapy, radiotherapy was initiated within 6 weeks after the end of chemotherapy, allowing both endocrine therapy and radiotherapy to be performed simultaneously. The clinical standard treatment regimen (chemotherapy, endocrine therapy, etc.) was developed based on postoperative pathological and immunohistochemical reports.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥55 years old；
2. Cytology or histology confirmed invasive breast cancer or intraductal carcinoma in situ (DCIS) with a clinical stage of Tis-1N0M0；
3. Patients who are willing to preserve milk and intend to undergo breast-conserving surgery；
4. If invasive breast cancer is confirmed, the surgical margin negative ≥2mm should be met. If DCIS is confirmed, the surgical margin should be negative ≥3mm；
5. ER≥ 30% and PR≥ 1%, HER2 negative；
6. Voluntary participation in this study, signed informed consent, good compliance, cooperate with follow-up.

Exclusion Criteria:

1. Simultaneous diagnosis of bilateral or multifocal breast cancer；
2. Previous ipsilateral breast cancer and/or prior chest wall radiation therapy；
3. There are active connective tissue diseases such as scleroderma and systemic lupus erythematosus in the chest；
4. The investigators did not consider the patient suitable for participation in any other conditions of the study.

Min Age: 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The clinical stage of Tis-1N0M0 in patients undergoing breast conserving surgery for early breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 620 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2026-11-19 (Estimated); Study Completion 2026-11-19 (Estimated)

PRIMARY OUTCOMES:
LRFS | At least 5 years
  There was no local recurrence survival

CONTACTS AND LOCATIONS:
Overall Officials: cuizhi GENG, archiater, Study Director — Hebei Medical University Fourth Hospital
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China